CLINICAL TRIAL: NCT01902927
Title: Modulation of Dyspnea Perception During Exercise in COPD Patients Using Attentional Distraction : a Pilot Study
Brief Title: Modulation of Dyspnea Perception During Exercise in COPD Patients Using Attentional Distraction
Acronym: DVD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Maltais, Francois, M.D. (Industry); Saey, Didier, M.D. (Individual); Dr Louis Laviolette (Unknown); Dr Thomas Similowski (Unknown)
Responsible Party: Principal Investigator, Philippe Gagnon, PhD Candidate, PhD, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple
Other Study IDs: DVD-20948
Record Dates: First submitted 2013-07-10; First posted 2013-07-18 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Exercise tolerance; Dyspnea; Affective distraction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- COPD patients (Experimental): COPD patients will perform a constant workrate treadmill exercise test until exhaustion with positve/neutral/negative visual distraction images during the exercise test assigned in a randomized order
  Interventions: Other: Attentional distraction using IAPS protocol (standardized images)

INTERVENTIONS:
Other: Attentional distraction using IAPS protocol (standardized images) — Positive, Negative and Neutral Attentional distraction will be presented using IAPS protocol (standardized images) during exercise tests

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major health problem whose prevalence is increasing rapidly. The gradual decrease in exercise tolerance is one of the usual consequences of COPD that affects the functional independence and quality of life of patients.

In COPD patients, breathlessness and muscle fatigue are the main symptoms limiting exercise. Recent studies have shown that most of the physiological mechanisms of psychological factors such as emotions, motivation, memory, personality, expectations, or prior experience can greatly influence and modulate the perception of breathlessness. It has been proposed that the attentional distraction (visual or auditory) during exercise may be associated with a decrease in anxiety and shortness of breath and could improve exercise tolerance in COPD. We therefore propose to study the impact of attentional strategies of distraction on the perception of dyspnea and walking tolerance in patients with COPD.

The research hypotheses are:

i) Compared with exposure to a strategy of negative attentional distraction during exercise, exposure to a strategy of positive attentional distraction will improve walking exercise tolerance in patients with COPD;

ii) For a given level of effort, sensory perception and emotional perception will be enhanced by exposure to a strategy of positive attentional distraction.

Ten subjects with moderate to severe COPD will be recruited at the Research Center of the Institut Universitaire de cardiologie et de pneumologie de Québec (CRIUCPQ). During an assessment visit, we will measure complete pulmonary function, body composition and maximal functional capacity during a maximal incremental test work performed on a treadmill.

During two subsequent experimental visits, and after spirometry control, participants will perform a walking test performed on a treadmill at an intensity corresponding to 75% of maximum effort during maximal incremental test. The test will be carried out in combination with a strategy of either positive attentional distraction, neutral attentional distraction or negative attentional distraction . The order of the condition will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history > 10 pack-years
* Post-BD FEV1 [30-80 % predicted value]
* Post-BD FEV1/FVC < 70 %
* Age [50-80 yrs]
* Voorips score < 9

Exclusion Criteria:

* Exacerbation < 4 weeks
* Asthma, Neoplasia, Cardiac failure, Diabetes
* Neuromuscular limitations
* Major depression or other psychiatric disorders
* BMI > 30 kg/m2
* PaO2 < 60 mmHg or oxygenotherapy
* Involvement in a structured and regular physical activity program

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance | During each experimental visit (V2-V3-V4), from the start to the end of the exercise test (limited by symptoms of the patients). Participants will be followed for an expected period of 3 weeks (from date of randomization to the completion of the study)
  The exercise tolerance (sec) will be defined as the time to exhaustion following a standardized constant workrate treadmill walking test corresponding to 75 % of maximal workload previously determined.

SECONDARY OUTCOMES:
Dyspnea perception | During visit 2-3-4, from start to end of the endurance exercise test at every 90-sec intervals, up to 20 minutes. Participants will be followed for an expected period of 3 weeks (from date of randomization to the completion of the study)
  The dyspnea intensity will be measured using a 10-point Borg scale during the exercise test
Dyspnea affective perception | During visit 2-3-4, from start to end of the endurance exercise test at every 90-sec intervals, up to 20 minutes. Participants will be followed for an expected period of 3 weeks (from date of randomization to the completion of the study)
  The affective perception of dyspnea will be measured using the mutlidimensionnal dyspnea profile questionnaire (MDP), graded on a 10-point scale

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Centre de recherche - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ)
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec, Canada